CLINICAL TRIAL: NCT01809405
Title: Validation of Sexual Function Scale in Female Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Yoon Park, Senior researcher, National Cancer Center, Korea
Other Study IDs: NCCNCS-12-685
Record Dates: First submitted 2013-03-02; First posted 2013-03-12 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Sexuality; Cancer; Healthy Women
MeSH Terms: conditions — Sexuality; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
To validate the FSFI(Female Sexual Function Index)-K, FSFI - 6 item and Quality of Sexual Function(QSF) version in Korean language of the cancer patients.

DETAILED DESCRIPTION:
Due to the observational nature of the study which aims to evaluate the internal consistency and validity of the Korean version of Questionnaire, formal sample size and power calculations were not performed. When the number of observations (items) per subject ranges from 4 to 6, roughly 152-199 patients are required to show 10% increase in intraclass correlation from baseline ICC of 30% with 85% power and 5% type I error rate. The sample size was determined based on this calculation and practical considerations.

The pilot study will be performed based on 30 people (include reference), and the main study will include 1100 people (considering 10% drop-out from 200 people in each group) cancer type (ovary, cervix, endometrium, and breast) and healthy female. Total 1130 patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women

  * Female without history of cancer
  * Cancer free as of the most recent linkage
  * At least 18 years of age
  * Able to speak and read Korean
  * Sexual activity within 3months.
* Female cancer patient

  * History of gynecological or breast cancer
  * At least 18 years of age
  * Able to speak and read Korean
  * Sexual activity within 3months.

Exclusion Criteria:

* Women who are unable to complete the questionnaires.
* Refuse to participate in the survey.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 1130 adult women living in Korea
Sampling Method: Probability Sample
Enrollment: 1130 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
sexuality | 2-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea